CLINICAL TRIAL: NCT02021552
Title: Genetic Polymorphisms & The Risk for Sepsis After Trauma
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Grant E. O'Keefe, Professor, University of Washington
Other Study IDs: 44109-A
Record Dates: First submitted 2013-12-09; First posted 2013-12-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Trauma
Keywords: Trauma; Sepsis
MeSH Terms: conditions — Wounds and Injuries; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White blood cells extracted from discarded blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- trauma patients: trauma patients 18 years or older requiring treatment in the ICU >24 hours. All subjects will undergo blood sampling.
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — 5 ml blood sampling

SUMMARY:
The specific aim of this is to establish a cohort of severely injured patients admitted to our trauma center. Investigators will collect DNA, utilizing discarded blood samples, from 3000 injury victims in an effort to identify perhaps 50 - 100 single-nucleotide polymorphisms (SNP) (out of 1000s) that can be used, when taken together, to identify patients at highest risk for developing complicated sepsis and death.

DETAILED DESCRIPTION:
The specific aim of this is to establish a cohort of severely injured patients admitted to our trauma center. Investigators will collect DNA, utilizing discarded blood samples, from 3000 injury victims in an effort to identify perhaps 50 - 100 single-nucleotide polymorphisms (SNP) (out of 1000s) that can be used, when taken together, to identify patients at highest risk for developing complicated sepsis and death

ELIGIBILITY:
Inclusion Criteria:

Admitted to the Intensive Care Unit (ICU) at Harborview Medical Center after suffering a traumatic injury

* ability to obtain a 5 ml blood sample
* Expected to be in the ICU for more than 24 hours

Exclusion Criteria:

* We will exclude subjects with chronic medical conditions for the reasons stated above as well as vulnerable populations (children, pregnant females, and prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort in which patients with severe injury, defined by combined anatomic injuries sufficient to require admission to the intensive care unit for treatment (blood transfusions, mechanical support of respiration) and intensive monitoring that is expected to be required for more than 24 hours, will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Investigators aim to identify up to 100 single-nucleotide polymorphisms (out of 1000s) that can be used, when taken together, to identify patients at highest risk for developing complicated sepsis and death. | 3 years
  The investigators will be studying whether baseline genetic difference can be used in the future to identify patients at high risk and conversely those at low risk for complicated post-traumatic infections.

CONTACTS AND LOCATIONS:
Overall Officials: Grant O'Keefe, MD, Principal Investigator — Professor; Dept of Surgery
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified samples and data will be available to other investigators at the discretion of the Principal Investigator.